CLINICAL TRIAL: NCT01750931
Title: AN OPEN LABEL, BALANCED, RANDOMIZED, TWO-TREATMENT, TWO-PERIOD, TWO-SEQUENCE, CROSSOVER, SINGLE ORAL DOSE, BIOEQUIVALENCE STUDY OF MELOXICAM GSK 15 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND MOBIC® 15 MG TABLETS OF BOEHRINGER INGELHEIM PHARMA GMBH & CO. KG BINGER STR.173, 5521 INGELHEIM AM RHEIN, GERMANY, IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FED CONDITION.
Brief Title: This Study is Randomised, Single Oral Dose Bioequivalence Study of Meloxicam GSK 15 MG Tablets.
Acronym: BA/BE: 250/12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117176
Record Dates: First submitted 2012-11-28; First posted 2012-12-17 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: BE study of Meloxicam GSK 15mg
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meloxicam GSK 15mg (Other): A randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study under fed condition
  Interventions: Drug: Meloxicam GSK 15mg; Drug: Mobic 15mg
- Mobic 15mg (Other): A randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study under fed condition
  Interventions: Drug: Meloxicam GSK 15mg; Drug: Mobic 15mg

INTERVENTIONS:
Drug: Meloxicam GSK 15mg — To demonstrate the bioequivalence of Meloxicam 15 mg tablets manufactured by Savipharm J.S.C, Vietnam and Mobic® 15 mg tablets of Boehringer Ingelheim Pharma GmbH & Co.KG Binger Str.173, 5521 Ingelheim am Rhein, Germany, in healthy adult human male subjects under fed condition
Drug: Mobic 15mg — To demonstrate the bioequivalence of Meloxicam 15 mg tablets manufactured by Savipharm J.S.C, Vietnam and Mobic® 15 mg tablets of Boehringer Ingelheim Pharma GmbH & Co.KG Binger Str.173, 5521 Ingelheim am Rhein, Germany, in healthy adult human male subjects under fed condition

SUMMARY:
It is a randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study of Meloxicam GSK 15 mg tablets manufactured by Savipharm J.S.Cc, Vietnam and Mobic® 15 mg tablets of Boehringer Ingelheim Pharma GmbH & Co. KG Binger Str.173, 5521 Ingelheim am Rhein, Germany, in healthy, adult, human male subjects under fed condition. It is a pivotal study to demonstrate the bioequivalence of Meloxicam GSK 15 mg tablets manufactured by Savipharm J.S.C, Vietnam and Mobic® 15 mg tablets of Boehringer Ingelheim Pharma GmbH & Co.KG Binger Str.173, 5521 Ingelheim am Rhein, Germany, in healthy adult human male subjects under fed condition.

This study will enroll 28 healthy adult human male subjects

DETAILED DESCRIPTION:
The objectives of this study are to:

To demonstrate the bioequivalence of Meloxicam GSK 15 mg tablets manufactured by Savipharm J.S.C, Vietnam and Mobic® 15 mg tablets of Boehringer Ingelheim Pharma GmbH & Co.KG Binger Str.173, 5521 Ingelheim am Rhein, Germany, in healthy adult human male subjects under fed condition To monitor the safety of the study subjects. Study design: A randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study under fed condition. It is a pivotal study Sample size estimation: Based on the literature available [Public assesment report Scientific Discussion Meloxicam "Arrow" Tablets 7.5 and 15 mg Meloxicam, DK/H/0905/001-002/MR] sample size of 28 subjects will be enough to meet the study objective. And 28 healthy adult human male subjects will be enrolled.

Screening procedures:

Demographic data, medical and medication histories, complete physical examination, height, weight and BMI as well as 12 lead ECG, chest X-ray [PA view], vital signs [blood pressure, pulse rate, respiratory rate and oral temperature], hematology, biochemistry, HIV1& 2, Hepatitis B and C, RPR test for Syphilis and urine analysis will be done at screening.

Urine drug screen, Liver chemistry test and Breath alcohol test to be done prior to each check-in.

Breath alcohol test to be done prior to each ambulatory visit blood collection. Housing: The study subjects will be housed at least 11 h prior to drug administration until after the 24 h blood sampling in each study period. The housing will be followed by three ambulatory visits [48, 72 and 96 hr post dose] during each period.

Study Meals Supervised fast for at least 10 h before dosing day breakfast will be maintained in each period. High calorie high fat breakfast will be served to subjects to start to consum 30 minutes before the scheduled dosing time. After dosing lunch, snacks and dinner will be served at 5, 8 and 12 h respectively. Meal plans will be identical for both the study periods.

Water will be permitted ad libitum except for 1 h before and until 1 h after post-dose.

Drug Administration:

As per the randomization schedule, one tablet of either test or reference product will be orally administered to each subject in each period in sitting posture, at 30 minutes after start of consuming served high calorie high fat breakfast on an overnight fast of at least 10 h. The investigational products will be administered with 240 ± 2 mL of water.

Subjects will be instructed not to chew or crush the tablet but should be swallowed. Compliance for dosing will be assessed by identification of subjects with subject ID card, identification of label on investigational product to confirm correct allocation of treatment and checking the oral cavity immediately after dosing.

Restrictions Subjects will remain in upright position [sitting or ambulatory] for two hours after dosing in each period except when clinically indicated to change the posture. The subjects will fast for at least 10 h prior to dosing day breakfast and 5 h post-dose. Water will be permitted ad libitum except for 1 h before and until 1 h after post dose.

Blood sampling:

In each period of the study, 26 blood samples of 6 mL each will be collected in K2EDTA vacutainers via an indwelling catheter placed in one of the forearm veins. Heparin-lock technique will be used to prevent clotting of blood in the indwelling catheter. Before each in-house blood sample is drawn through catheter, 0.5 mL of blood will be discarded so as to purge the heparin containing blood sample in the catheter. Blood can also be collected by direct venipuncture in case of cannula blockage, during ambulatory visits or for any other practical reasons. The two pre-dose blood samples will be collected within a period of 1 h before the drug administration. The post-dose blood samples will be collected at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 16.0, 24.0, 48.0, 72.0 and 96.0 h. The 48.0, 72.0 and 96.0 h post dose blood samples will be collected during ambulatory visits by direct venipuncture. Immediately after collection of blood, the sample will be kept in ice bath. After collecting the blood samples from all the subjects at each sampling time point, samples will be centrifuged at 4oC with 3500 rpm for 10 minutes. The plasma samples will be separated in duplicate and stored in pre-labeled polypropylene tubes at -70 ± 10°C or colder pending assay. The time interval between sample collection and the start of centrifugation should not exceed more than 45 minutes.

The total volume of blood drawn including the volume necessary for the laboratory tests, PK sample analysis and the volume of blood discarded before each in house blood draw will be about 360 mL per subject for the entire study.

Washout Period: Washout period will be of at least 14 days, but not exceeding 21 days between two dosing days.

Pharmacokinetic Parameter: Cmax, Tmax, AUC0-t, AUC0-∞, AUC%_Extrap, Kel and t1/2 Analytical Methods: Meloxicam in plasma will be estimated using validated LC-MS/MS method.

Statistical Methods: Statistical analyses will be done using SAS® version 9.2 or higher. Analysis of variance [ANOVA] for log-transformed pharmacokinetic parameters [Cmax, AUC0-t and AUC0-∞] and two one-sided tests [Schuirmann] for bioequivalence will be performed. Power, ratio and 90% confidence interval for log-transformed pharmacokinetic parameters - Cmax, AUC0-t and AUC0-∞ will be calculated.

Standards for Bioequivalence: The calculated 90% Confidence Interval for the test to reference ratio of Meloxicam should fall within the range of 80%-125% for log transformed Cmax, AUC0-t and AUC0-∞ for the conclusion of bioequivalence.

Adverse Events The investigator or site staff is responsible for detecting, documenting and reporting events that meet the definition of an AE or SAE.

AEs will be collected from the start of Study Treatment and until the follow-up contact. Medical occurrences that begin prior to the start of study treatment but after obtaining informed consent may be recorded on the Medical History/Current Medical Conditions CRF.

SAEs will be collected over the same time period as stated above for AEs. However, any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact. All SAEs will be recorded and reported to the sponsor within 24 hours.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he considers the event reasonably related to the study treatment or study participation, the investigator would promptly notify the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male human subjects within the age range of 18 to 45 years inclusive.
* Heght not less than 50 kg.
* Normal BMI [18.5 to 24.99 kg/m2 inclusive].
* Willingness and capability to provide written informed consent to participate in the study.
* Free of significant diseases or clinically significant abnormal findings based on medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
* Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* ECG normal for morphology and measurements. QTcB or QTcF < 450 msec or QTc < 480 msec in subjects with Bundle Branch Block, based on an average from three ECGs obtained over a brief recording period.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed below. This criterion must be followed from the time of the first dose of study medication until one week of last dose administration.
* Condom plus partner use of a highly effective contraceptive such as occlusive cap (diaphragm or cervical/vault cap) plus spermicidal agent (foam/gel/film/cream/suppository), oral contraceptive, injectable progesterone, implant of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, or intrauterine device.

OR

* Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* History or presence of significant: Cardiovascular, pulmonary, hepatic, renal, hematological, gastro-intestinal, endocrine, immunologic, dermatologic, neurological, psychiatric disease.
* History or presence of significant:
* Alcohol dependence or alcohol abuse during past one year.
* Drug abuse [Marijuana [THC], Cocaine, Morphine, Benzodiazepines, Barbiturates and Amphetamine] for the last 6 months.
* Smoking of more than 5 cigarettes per day or consumption of other forms of tobacco containing products.
* Asthma, urticaria or other allergic type reactions after taking aspirin or any other drug.
* Ulceration or history of gastric and / or duodenal ulcer.
* Jaundice in the past 6 months.
* Bleeding disorder.
* Allergy to the test drug or any drug chemically similar to the drug or to the excipients of the products under investigation.
* Donation of 500 mL or more blood within 8 weeks prior to receiving the first dose of study drug.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Any difficulty in accessibility of forearm veins for cannulation or blood sampling.
* Refusal to consume high calorie high fat breakfast 30 minutes before scheduled dosing time and abstain from food for at least 5 h post dose in each period.
* Refusal to abstain from fluid for at least 1 h prior to and 1 h post each dose.
* Positive breath alcohol test result found on the day of check-in.
* Positive urine test result for drug of abuse found on the day of check-in.
* History of difficulty in swallowing tablet.
* Use of any concomitant medication [including over-the-counter products, vitamins etc.] for 14 days preceding the study drug administration.
* Use of drugs which induce or inhibit metabolizing enzymes within 30 days prior to receiving the first dose of study medication.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-09-12 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 28 participants were enrolled from September-2013 to October-2013. At each study period participants received test (GlaxoSmithKline [GSK]-meloxicam 15 milligram [mg] tablet) and reference (Mobic®-meloxicam 15 mg tablet) products. Mobic is registered product of Boehringer Ingelheim Pharma GmbH and Company, Germany.
Groups:
- GSK-meloxicam Then Mobic-meloxicam: In this period of the study, participants received a single oral dose of test (GSK-meloxicam 15 mg tablet) followed by reference (Mobic-meloxicam 15 mg tablet) product as per the randomization schedule with 240 milliliters (mL) of water 30 minutes after start of consumption of high fat high calorie breakfast on an overnight fast of at least 10 hours. Dosing was scheduled at specific intervals between 08:30 ante meridiem (am) to 08:56 am in each study period. A washout period of 14 days was maintained between the dosing of each period.
- Mobic-meloxicam Then GSK-meloxicam: In this period of the study, participants received a single oral dose of reference (Mobic-meloxicam 15 mg tablet) followed by test (GSK-meloxicam 15 mg tablet) product as per the randomization schedule with 240 milliliters (mL) of water 30 minutes after start of consumption of high fat high calorie breakfast on an overnight fast of at least 10 hours. Dosing was scheduled at specific intervals between 08:30 ante meridiem (am) to 08:56 am in each study period. A washout period of 14 days was maintained between the dosing of each period.
Period: Period 1
Arm/Group | GSK-meloxicam Then Mobic-meloxicam | Mobic-meloxicam Then GSK-meloxicam
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Wash Out
Arm/Group | GSK-meloxicam Then Mobic-meloxicam | Mobic-meloxicam Then GSK-meloxicam
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | GSK-meloxicam Then Mobic-meloxicam | Mobic-meloxicam Then GSK-meloxicam
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK-meloxicam 15 mg + Mobic-meloxicam 15 mg: In each period of the study, participants received a single oral dose of test (GSK-meloxicam 15 mg tablet) or reference (Mobic-meloxicam 15 mg tablet) product as per the randomization schedule with 240 mL of water 30 minutes after start of consumption of high fat high calorie breakfast on an overnight fast of at least 10 hours. Dosing was scheduled at specific intervals between 08:30 am to 08:56 am in each study period. A washout period of 14 days was maintained between the dosing of each period.
Arm/Group | GSK-meloxicam 15 mg + Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 25.04 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Region of Enrollment [Number; unit: Participants]
  India | 28

OUTCOME MEASURES:

1. Primary Outcome: Maximum Drug Concentration During the Selected Dosing Interval (Cmax) After a Single Dose
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at indicated time points of each treatment period. The Cmax was taken directly from the plasma concentration-time profile of individual participants
Time Frame: Pre-dose (two samples collected within a period of 1 hour) and 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 5.5, 6.0, 6.5, 7.0, 7.5, 8.0, 9.0, 10.0, 12.0, 16.0, 24.0, 48.0, 72.0 and 96.0 hours post-dose in each treatment period
Population: All subject population: all participants who complete all periods of the study. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Groups:
- GSK-meloxicam 15 mg: In each period of the study, participants received a single oral dose of test product (GSK-meloxicam 15 mg tablet) as per the randomization schedule with 240 mL of water 30 minutes after start of consumption of high fat high calorie breakfast on an overnight fast of at least 10 hours. Dosing was scheduled at specific intervals between 08:30 am to 08:56 am in each study period.
- Mobic-meloxicam 15 mg: In each period of the study, participants received a single oral dose of reference (Mobic-meloxicam 15 mg tablet) as per the randomization schedule with 240 mL of water 30 minutes after start of consumption of high fat high calorie breakfast on an overnight fast of at least 10 hours. Dosing was scheduled at specific intervals between 08:30 am to 08:56 am in each study period.
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Nanogram per milliliter | 1889.579 (15.31) | 1844.423 (15.74)
Statistical Analysis 1: Comparison: GSK-meloxicam 15 mg vs Mobic-meloxicam 15 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; p = 0.4396, ANOVA; Percent ratio = 102.45, 95% CI 2-sided [99.40 to 105.59]

2. Primary Outcome: Time to Maximum Concentration (T-max)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. The Tmax was taken directly from the plasma concentration-time profile of individual participants. Plasma samples for PK analysis were drawn at indicated time points.
Time Frame: as for outcome 1
Population: All subject population
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Hour | 5.50 (16.0) [5.00 to 8.02] | 5.50 (14.7) [5.00 to 8.00]

3. Primary Outcome: The Area Under the Plasma Concentration Versus Time Curve (AUC) After a Single Dose
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. AUC(0-t) was area under the plasma concentration-time curve from time of administration until the time of last quantifiable concentration. The area under the plasma concentration-time curve (AUC0-infinity), was estimated by linear trapezoidal rule and was sum of the AUC0-t and extrapolated to infinity by dividing the estimated last measurable plasma concentration by elimination rate constant lambda z. Where lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data after each single dose. The AUC0-infinity was the sum of the estimated and extrapolated parts.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram.hour per milliliter
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Nanogram.hour per milliliter
  AUC(0-t) | 57499.339 (31.00) | 54750.590 (33.21)
  AUC(0-inf) | 62687.372 (44.49) | 61269.334 (50.30)
Statistical Analysis 1: Comparison: GSK-meloxicam 15 mg vs Mobic-meloxicam 15 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; p = 0.9712, ANOVA; Percent ratio = 105.02, 95% CI 2-sided [99.69 to 110.63] — Comparison of AUC0-t between group GSK-meloxicam 15 mg and Mobic-meloxicam 15 mg
Statistical Analysis 2: Comparison: GSK-meloxicam 15 mg vs Mobic-meloxicam 15 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; p = 0.9951, ANOVA; Percent ratio = 102.31, 95% CI 2-sided [99.05 to 105.69] — Comparison of AUC0-infinity between group GSK-meloxicam 15 mg and Mobic-meloxicam 15 mg

4. Primary Outcome: The Percentage of Area Under Curve Extrapolated to Arrive at AUC0-infinity (AUCpercentage [%]_Extrap [Residual Area]) After a Single Dose
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. The percentage of area under curve extrapolated to arrive at AUC0-infinity (AUC%_Extrap [residual area]) was determined by AUC0-infinity minus AUC0-t divided by AUC0-infinity multiplied by 100.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC Extrapolated
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Percentage of AUC Extrapolated | 4.32 (119.8) | 5.02 (132.1)

5. Primary Outcome: Elimination Rate Constant (Kel) After a Single Dose
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. The apparent first-order elimination or terminal rate constant was calculated from a semilogarithmic plot of the plasma concentration versus time. The parameter was calculated by linear least-square regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Per hour | 0.032 (33.91) | 0.030 (34.50)

6. Primary Outcome: Elimination Half Life (T-half) After a Single Dose
Description: The T-half was calculated using the following formula by dividing 0.693 (natural logarithm of 2) with lambda z, where lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data after each single dose.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Median (Full Range); unit: Per hour
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Per hour | 21.362 [11.437 to 66.697] | 22.337 [12.522 to 92.217]

7. Secondary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, is medically important event or reaction, is associated with liver injury Alanine amino transferase (more than equal to [>=] 3 fold upper normal of limit [ULN]) or total bilirubin (>=2 fold ULN) or international normalization ratio more than 1.5. Refer to the general AE/SAE module for a list of AEs and SAEs.
Time Frame: Up to 20 days
Population: All subject population.
Measure: Number; unit: Participants
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
Number analyzed (Participants) | 28 | 28
Participants
  Any AE | 0 | 1
  Any SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: AE and SAE were reported through out the study (up to 20 days)
Description: For reporting AE and SAE, all subject population was used.
Arm/Group | GSK-meloxicam 15 mg | Mobic-meloxicam 15 mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK-meloxicam 15 mg (N=28) | Mobic-meloxicam 15 mg (N=28)
Headache (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.